CLINICAL TRIAL: NCT03222466
Title: A Randomized Trial to Assess Whether Co-creating Patient Educational Materials With Patients Has Added Value Over Researchers and Clinicians Developing Patient Education Materials and Engaging Patients During Usability Testing Only.
Brief Title: Patient Educational Materials for Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SMH REB #:16-376
Record Dates: First submitted 2017-07-11; First posted 2017-07-19 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Patient Educational Materials
Keywords: Patient educational materials; prostate cancer; co-creation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-created PEM (Experimental): A co-created PEM has been designed in collaboration with patients. Participants receiving the intervention will be asked to read and answer questions before and after viewing the co-created PEM.
  Interventions: Other: Co-created PEM
- Traditional PEM (No Intervention): Participants will be asked to read and answer questions before and after viewing the traditional PEM created by clinicians and researchers.

INTERVENTIONS:
Other: Co-created PEM — A co-created PEM has been designed in collaboration with patients.
  Arms: Co-created PEM

SUMMARY:
Although the harms of screening for prostate cancer with the prostate-specific antigen (PSA) test outweigh the benefits, 560,000 Ontario men undergo PSA screening each year. Guideline developers, such as the Canadian Task Force on Preventive Health Care (CTFPHC), have disseminated patient educational materials (PEMs) on PSA screening widely in Ontario, yet men remain confused about screening harms and benefits. One potential contributing factor may be that PEMs are typically developed by researchers and clinicians and may not address patient barriers to change. The investigators will assess whether a PSA screening PEM that is co-created with patients provides added value over PEMs developed using the traditional approach (i.e., researchers and clinicians develop a PEM with patient involvement in usability testing only. The investigators will also assess satisfaction with the engagement process and calculate the costs and resources required for each method (i.e. co-creation, usability, and recommendations only). This study will generate a PSA screening PEM to help patients make evidence-based screening decisions. It will also help Ontario organizations, including Cancer Care Ontario, identify optimal methods for developing PEMs for PSA screening and other areas of preventive health care, such as breast and colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking men aged 40+ years will be eligible to take part in the project if they have never been diagnosed with prostate cancer and do not have any signs or symptoms of prostate cancer.

Exclusion Criteria:

* Individuals will not be eligible for the project if they indicate that they are a health care professional or have any conflicts of interest relevant to the guideline topic (e.g., owning shares in a company related to prostate cancer treatment).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 573 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Pretest-posttest change in prostate cancer screening decisional conflict and intention to be screened between the co-created PEM group and the traditional PEM group. | This measure will be assessed from date of randomization until date of survey completion, assessed up to 1 month.
  The investigators will assess differences and changes in prostate cancer screening decisional conflict and intention to be screened for the co-created PEM group and the traditional PEM group using repeated measures ANOVAs.

SECONDARY OUTCOMES:
Pretest-posttest change in knowledge of prostate cancer screening | This measure will be assessed from date of randomization until date of survey completion, assessed up to 1 month.
  The investigators will assess the differences in the pretest-posttest change in prostate cancer screening knowledge between the co-created PEM group and the traditional PEM group using a 7-item knowledge measure. Assessed by conducting a repeated measures analysis of variance (ANOVA).
Comparison of PEM usability | This measure will be assessed from date of randomization until date of survey completion, assessed up to 1 month.
  The investigators will assess the differences between the two study arms in PEM/recommendation usability using a one-way ANOVA
Participant preference of PEM | This measure will be assessed from date of randomization until date of survey completion, assessed up to 1 month
  The investigators will evaluate participants' preferred material (co-created or traditional PEM). Use a chi-square test to analyze the difference in the proportion of patients who prefer each type of material.
Resources use for PEM development | This measure will be assessed after the intervention (survey) is administered (i.e., post analysis), up to 1 month.
  The investigators will record the resources required (e.g., personnel hours and participant reimbursement) for a health care organization to develop a co-created PEM in comparison to a PEM created by clinicians and researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No